CLINICAL TRIAL: NCT00643526
Title: An Open-Label, Randomized, Validation Study to Establish That the Design, Functionality, and Ergonomic Features of the Autoinjector Conform to Defined User Needs and Intended Use for Self-Administration by Subjects With Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, or Psoriasis
Brief Title: A Study to Test the Design, Functionality, and Ergonomic Features of the Autoinjector
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR014914
Record Dates: First submitted 2008-02-22; First posted 2008-03-26 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Psoriasis
Keywords: Rheumatoid arthritis; Psoriatic arthritis; Ankylosing spondylitis; Psoriasis; Autoinjector
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection Site: First Thigh Then Abdomen (Experimental): Participants will self inject subcutaneously placebo using auto injector at thigh followed by self injection of placebo subcutaneously at abdomen on Day 1.
  Interventions: Device: Pre-filled Auto-injector Containing Placebo
- Injection Site: First Abdomen then Thigh (Experimental): Participants will self inject subcutaneously placebo using auto injector at abdomen followed by self injection of placebo subcutaneously at thigh on Day 1.
  Interventions: Device: Pre-filled Auto-injector Containing Placebo

INTERVENTIONS:
Device: Pre-filled Auto-injector Containing Placebo — Participants will self-inject placebo subcutaneously at thigh and abdomen.

SUMMARY:
The main purpose of this study is to evaluate how well the autoinjector works in a group of people who are likely to use the autoinjector for injecting their medicine in the future. However, no active medicine is given by the autoinjector.

DETAILED DESCRIPTION:
This device (called an autoinjector) automatically injects medicine under the skin with a sterile needle, and is similar to other types of autoinjectors currently being used for this purpose. This trial has been designed to make sure that people, who are likely to use this device, are able to self-inject and understand the training material. A total of 68 subjects took part in the study. About half (30 patients) will have either Rheumatoid Arthritis (RA), psoriatic arthritis (PsA) or ankylosing spondylitis (AS) and the other half will have psoriasis (a type of skin disease), since this device will be used by patients with one of these diseases to inject their medication. The study is designed to have each patient complete 2 self-injections with the autoinjector in 2 different sites-one in the front of the thigh and one in the abdomen 2 inches away from the navel. The order of the first injection location is decided by randomization. The patient will have an equal chance of having the thigh or the abdomen as the first injection. The study staff will assess the subject's safety prior to the patient leaving the clinic. Two prefilled, 1mL placebo autoinjectors for subcutaneous injection

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to understand and sign an informed consent form
* Have one of the following diagnoses: rheumatoid arthritis/psoriatic arthritis/ankylosing spondylitis, or psoriasis
* Be willing and able to self-inject

Exclusion Criteria:

* Have a recent history of (within 6 months prior to study entry) or current diagnosis of a major bleeding or coagulation disorder
* Have a prior history of a inability to use an autoinjector
* Have an allergy to latex or any component of the autoinjector
* Female participants who are pregnant
* Are unwilling to complete the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To establish that the autoinjector, as designed, meets defined user needs and intended use for self administration by patients with RA, PsA, AS, and psoriasis | Day 1

SECONDARY OUTCOMES:
•To establish that the specific training, including the instructional video and the Instructions for Use, are appropriate, easy to understand, and able to be followed and implemented by patients with RA, PsA, AS, and psoriasis. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (2):
- United States (2):
  - Miami, Florida
  - Duncansville, Pennsylvania